CLINICAL TRIAL: NCT01537939
Title: ASUKI Step Pedometer Worksite Intervention
Acronym: ASUKI-Step
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Barbara E. Ainsworth, Professor, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ASUKI2009
Record Dates: First submitted 2012-02-18; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Physical Activity
Keywords: Physical Activity; Walking; Pedometer; Body Composition; Aerobic Fitness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Walking (Other): Quasi-experimental design with one-group, post-test only
  Interventions: Behavioral: ASUKI Step Worksite Pedometer Intervention

INTERVENTIONS:
Behavioral: ASUKI Step Worksite Pedometer Intervention — The intervention required participants to accumulate 10,000 steps each day for six months, with a 3-month follow-up period. Steps were recorded onto a study-specific website. Participants completed a website-delivered questionnaire four times to identify socio-demographic, health, psychosocial and environmental correlates of study participation. One person from each team at each university location was randomly selected to complete physical fitness testing to determine their anthropometric and cardiovascular health and to wear an accelerometer for one week.
  Other Names: Pedometer-monitored daily walking

SUMMARY:
ASUKI Step is designed to increase the number of days employees walk 10,000 steps and to reduce the number of days employees spend being inactive.

Study aims were:

1. to have a minimum of 400 employee participants from each university site reach a level of 10, 000 steps per day on at least 100 days (3.5 months) during the trial period;
2. to have 70% of the employee participants from each university site maintain two or fewer inactive days per week, defined as a level of less than 3,000 steps per day;
3. to describe the socio-demographic, psychosocial, environmental and health-related determinants of success in the intervention; and
4. to evaluate the effects of a pedometer-based walking intervention in a university setting on changes in self-perceived health and stress level, sleep patterns, anthropometric measures and fitness.

DETAILED DESCRIPTION:
ASUKI Step is a 9-month pedometer-based worksite intervention conducted at the Karolinska Institutet (KI) in Stockholm, Sweden and Arizona State University (ASU) in the greater Phoenix area, Arizona. ASUKI Step used a quasi-experimental design based on the theory of social support. Participants included 2,118 faculty, staff, and graduate students from ASU (n = 712) and KI (n = 1,406) who participated in teams of 3-4 persons. The intervention required participants to accumulate 10,000 steps each day for six months, with a 3-month follow-up period. Steps were recorded onto a study-specific website. Participants completed a website-delivered questionnaire four times to identify socio-demographic, health, psychosocial and environmental correlates of study participation. One person from each team at each university location was randomly selected to complete physical fitness testing to determine their anthropometric and cardiovascular health and to wear an accelerometer for one week. Incentives were given for compliance to the study protocol that included weekly raffles for participation prizes and a grand finale trip to Arizona or Sweden for teams with most days over 10,000 steps.

ELIGIBILITY:
Inclusion Criteria:

* Employed at Arizona State University (ASU)or the Karolinska Institute (KI)
* The ability to read, speak and understand English (ASU only)
* Not currently pregnant or lactating
* Free of physical problems that affect the ability to walk, and e) ages 18 and older

Exclusion Criteria:

* Inability to walk
* Not employed or a graduate student at ASU or the KI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2018 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Percent of sample walking 10,000 steps per day on at least 100 days (3.5 months) during the trial period. | End of walking intervention at 6 months
  Tally of the participants recording 10,000 steps on their pedometer log for 100 days of the 6 month walking intervention.

SECONDARY OUTCOMES:
Changes in self-perceived health and stress level, sleep patterns, anthropometric measures and fitness. | End of the 6 month walking study
  Compare the measures between the first week and the last week of the 6-month intervention study

CONTACTS AND LOCATIONS:
Overall Officials: Barbara E. Ainsworth, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Arizona State University and Karolinska Institutet, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Ainsworth BE, Der Ananian C, Soroush A, Walker J, Swan P, Poortvliet E, Yngve A. "ASUKI Step" pedometer intervention in university staff: rationale and design. BMC Public Health. 2012 Aug 15;12:657. doi: 10.1186/1471-2458-12-657. PMID 22894138